CLINICAL TRIAL: NCT06433557
Title: A Phase 2, Open-Label, Single-Arm, 156-week Trial to Investigate the Efficacy, Safety and Tolerability of Combined Once Weekly Navepegritide and Lonapegsomatropin in Children With Achondroplasia
Brief Title: A Phase 2 Clinical Trial to Evaluate Efficacy, Safety, and Tolerability of Navepegritide in Combination With Lonapegsomatropin in Children With Achondroplasia
Acronym: COACH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ascendis Pharma Growth Disorders A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASND0042
Record Dates: First submitted 2024-05-23; First posted 2024-05-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination of Navepegritide and Lonapegsomatropin (Experimental)
  Interventions: Drug: Combination of Navepegritide and Lonapegsomatropin administered as two separate s.c. injections

INTERVENTIONS:
Drug: Combination of Navepegritide and Lonapegsomatropin administered as two separate s.c. injections — For navepegritide, a once weekly s.c. dose of 100 μg CNP/kg. For lonapegsomatropin, a once weekly s.c. dose of lonapegsomatropin 0.30 mg hGH/kg as starting dose. Treatment duration of up to 156 weeks.

SUMMARY:
This proof-of-concept trial is being conducted to evaluate the efficacy, safety and tolerability of combination treatment with navepegritide and lonapegsomatropin administered as separate subcutaneous (SC) injections once weekly in children with achondroplasia (ACH) aged 2 to 11 years.

ELIGIBILITY:
Inclusion Criteria:

1. Written, signed informed consent and/or assent (if applicable) by the parent(s) or legal representative(s) of the participant, and as required by the IRB/HREC/IEC.
2. Male or female between 2 to 11 years of age (inclusive) at the time of Visit 1.
3. Clinical diagnosis of ACH with genetic confirmation of heterozygote genotype present at Visit 1. Documentation of historic test results are acceptable for proof of diagnosis.
4. Able to stand without assistance.
5. Parent(s)/caregiver(s)/legal guardian(s) willing and able to administer weekly SC injections of IMP and comply with all protocol requirements.
6. At least 6 months of growth and disease history from TCC-NHS-01 or TCC-201 or comparable growth and disease history available from medical records.
7. No intracranial pathology as confirmed by brain MRI (historical MRI obtained within 2 years prior to screening allowable).

Exclusion Criteria:

1. Participation in any interventional clinical trial within three months prior to screening (except TCC-201 or ASND0039).
2. Closed epiphysis at screening.
3. History of or suspected hypersensitivity to the IMP or related products.
4. Findings on fundoscopy at screening consistent with intracranial hypertension, papilledema, or evidence of any other retinal disease for which GH therapy is contraindicated.
5. Have a growth disorder or medical condition other than ACH that results in short stature or abnormal growth such as severe ACH with developmental delay and acanthosis nigricans (SADDAN), hypochondroplasia, GHD, Turner syndrome, pseudoachondroplasia, inflammatory bowel disease, celiac disease, hypothyroidism, hyperthyroidism, pre-diabetes, or diabetes mellitus.
6. Have received any dose of prescription and/or investigational medications or device intended to affect stature, growth, or body proportionality at any time prior to screening.
7. Receiving concurrent treatment with any agent that might influence growth or interfere with GH secretion or action:

   1. Inhaled corticosteroid therapy at a dose of >400 µg/day of inhaled budesonide or equivalent for more than 28 consecutive days total over the course of 12 months prior to screening.
   2. Require, or anticipated to require, chronic (>4 weeks) or repeated treatment (more than twice/year and >3 weeks/year) with systemic corticosteroids during participation in the trial.
   3. Currently using or have used within 12 months prior to screening any sex steroids (for example estrogen), non-steroidal anabolic agents (for example, oxandrolone) or gonadotropin-releasing hormone (GnRH) analogues treatment.
   4. Treatment for attention-deficit hyperactive disorder (ADHD) such as methylphenidate.
8. Known history or presence of injury or disease of the growth plate(s), other than ACH, that affects growth potential of long bones.
9. Known history of any bone-related surgery affecting growth potential of long bones, such as Orthopaedic reconstructive surgery for bone lengthening (procedures for leg bowing such as 8-plate are not exclusionary).
10. Cervicomedullary decompression surgery within 6 months prior to Screening or with anticipated need for repeat decompression surgery during the time of the trial.
11. Evidence at screening consistent with severe cervicomedullary junction compression based on clinical and/or radiologic findings that indicate immediate surgical intervention is required.
12. Ventriculoperitoneal shunt and laminectomy with full recovery within 6 months prior to Screening.
13. Salter-Harris fracture within 6 months prior to screening (within 2 months for fracture of digits and buckle fractures).
14. Clinically significant musculoskeletal disease, such as Salter-Harris fractures or clinical and/or radiographic evidence of severe hip pathology.
15. Planned or expected surgical intervention during trial participation that may significantly affect trial parameters (confounding of safety events) or would prevent the participant from performing trial procedures. Minimally invasive surgeries such as insertion of grommets, adenoidectomy, tonsillectomy, or myringotomy tube placement, are permitted during the trial.
16. Severe untreated sleep apnoea or newly initiated sleep apnoea treatment (e.g., Continuous Positive Airway Pressure [CPAP] in the previous 2 months prior to screening).
17. Clinically significant finding or arrhythmia as determined by the investigator that indicates abnormal cardiac function or conduction that includes, but is not exclusive to:

    1. Repaired or unrepaired coarctation.
    2. Moderate or greater complexity congenital heart disease including tetralogy of Fallot, Atrioventricular septal defects, truncus arteriosus, total anomalous pulmonary venous return, double outlet right ventricle, or single ventricle heart disease.
18. QT corrected using Fridericia's correction (QTcF) ≥ 450 msec at screening.
19. Known history or presence of condition that impacts haemodynamic stability (such as autonomic dysfunction and orthostatic intolerance).
20. Known history or presence at screening of the following:

    1. Chronic anaemia (iron deficiency anaemia that is resolved or considered adequately treated in the Investigator's opinion is allowed).
    2. Chronic renal insufficiency defined as estimated glomerular filtration rate (eGFR) according to the revised bedside Schwartz equation less than <60 mL/min/1.73 m2 for >3 months.
    3. Chronic or recurrent illness that can affect hydration or volume status, including conditions associated with decreased nutritional intake or increased volume loss.
21. Known history or presence of malignant disease.
22. Hepatic transaminases (aspartate aminotransferase (AST) or alanine transferase (ALT)) greater than 3x upper limit of normal (ULN) at screening.
23. Serum 25-hydroxy-vitamin D (25OHD) level of <30 nmol/L (<12 ng/mL) at screening.

    Participants with 25OHD levels between 30-50 nmol/L (12-20 ng/mL) may be enrolled provided treatment with Vitamin D supplementation is initiated.
24. Any disease or condition that, in the opinion of the Investigator, may make the participant unlikely to fully complete the trial, may confound interpretation of trial results, or may present undue risk from receiving trial treatment. This could include family situations, complications or manifestations, or medications that might impact safety or be considered confounding.
25. Sexually active male and female participants who are unwilling or unable to use a highly effective form of contraception for the entire trial period and for 90 days after last dose of trial treatment.
26. Female participants who are pregnant, lactating or breastfeeding.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Annualized growth velocity | Week 52
  cm per year, compared to navepegritide alone
Treatment-emergent adverse events (TEAEs). | Throughout the trial for 156 weeks
  safety profile of navepegritide and lonapegsomatropin

SECONDARY OUTCOMES:
Annualized growth velocity | From start until 156 weeks
  cm per year

CONTACTS AND LOCATIONS:
Locations (3):
- Ascendis Pharma Investigational Site, Copenhagen, Denmark
- Ascendis Pharma Investigational Site, Dublin, Ireland
- Ascendis Pharma Investigational Site, London, United Kingdom